CLINICAL TRIAL: NCT00094666
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, 30-Night Polysomnographic Study of MK0928 in Elderly Patients With Primary Insomnia
Brief Title: Elderly Primary Insomnia Polysomnographic Study (0928-002)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-002; MK0928-002; 2004_085
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0928, gaboxadol / Duration of Treatment - 6 weeks
Drug: Comparator: placebo / Duration of Treatment - 6 weeks

SUMMARY:
The purpose of the study is to test the safety and effectiveness of an Investigational Drug on insomnia in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with a diagnosis of primary insomnia and in good physical and mental health

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 465
Dates: Start 2004-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Amount of time spent awake and time to fall asleep at night after two days

SECONDARY OUTCOMES:
Amount of time spent awake and time to fall asleep at night after 30 days
Amount of deep sleep after two days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Lankford DA, Corser BC, Zheng YP, Li Z, Snavely DB, Lines CR, Deacon S. Effect of gaboxadol on sleep in adult and elderly patients with primary insomnia: results from two randomized, placebo-controlled, 30-night polysomnography studies. Sleep. 2008 Oct;31(10):1359-70. PMID 18853933
- [Derived] Svetnik V, Snyder ES, Tao P, Roth T, Lines C, Herring WJ. How well can a large number of polysomnography sleep measures predict subjective sleep quality in insomnia patients? Sleep Med. 2020 Mar;67:137-146. doi: 10.1016/j.sleep.2019.08.020. Epub 2019 Sep 11. PMID 31926466